CLINICAL TRIAL: NCT01927757
Title: A Single Arm Trial to Evaluate the Efficacy of Etanercept in Moderate to Severe Rheumatoid Arthritis Patients Who Failed to Respond or Lost a Satisfactory Response to Treatment With Adalimumab When Used as Their First Biologic Agent
Brief Title: Evaluating Etanercept Use in Patients With Moderate to Severe Rheumatoid Arthritis Who Have Lost Response to Adalimumab
Acronym: ROCkIES
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Business decision due to slow enrollment
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20120125
Record Dates: First submitted 2013-06-05; First posted 2013-08-23 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Moderate to Severe Rheumatoid Arthritis
Keywords: rheumatoid arthritis; etanercept; arthritis; adalimumab failure to respond; loss of response to adalimumab; ACR20; methotrexate; Swollen joints; tender joints
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Etanercept; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etanercept (Experimental): Participants received etanercept 50 mg administered subcutaneously once a week with methotrexate for 24 weeks
  Interventions: Biological: Etanercept; Drug: Methotrexate

INTERVENTIONS:
Biological: Etanercept — Administered by subcutaneous injection
  Other Names: Enbrel®
Drug: Methotrexate — Background methotrexate at least 15 mg weekly

SUMMARY:
To evaluate the efficacy of etanercept in adults with moderate-to-severe rheumatoid arthritis (RA) who did not respond to or lost a satisfactory response to adalimumab when used as their first biologic agent.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Diagnosed with moderate to severe rheumatoid arthritis for at least 6 months
* Active RA with at least 3 swollen and tender joints
* Failure to respond to a combination treatment of adalimumab and methotrexate (must have taken combination at least 3 months) or loss of a satisfactory response to the combination of adalimumab and methotrexate, which was taken for at least 6 months (if currently taking adalimumab must complete 2 weeks without it prior to starting study drug)
* Negative for hepatitis B and C
* Negative serum and urine pregnancy tests before starting study
* currently taking (stable dose) 15 mg methotrexate weekly for at least 8 weeks/has been taking methotrexate for at least 12 weeks total - lower dose of 10 mg per week is permitted with documented intolerability
* Normal chest X-ray within 3 months
* Negative testing for tuberculosis (TB)

Exclusion Criteria:

* Class IV RA (wheel-chair or bed-bound)
* Significant concurrent medical conditions, including: (uncontrolled type 1 diabetes, poorly controlled type 2 diabetes, symptomatic heart failure, myocardial infarction in past year, history of unstable angina within past year, uncontrolled hypertension, severe chronic pulmonary disease, major chronic inflammatory or connective tissue disease other than RA, Multiple sclerosis, active malignancy, or history of cancer, alcoholic hepatitis or history of alcoholic liver disease)
* Other inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-05-06 (Actual); Primary Completion 2015-06-11 (Actual); Study Completion 2015-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (42):
- United States (32):
  - Research Site, Tuscaloosa, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Covina, California
  - Research Site, Hemet, California
  - Research Site, Murrieta, California
  - Research Site, San Diego, California
  - Research Site, Victorville, California
  - Research Site, Denver, Colorado
  - Research Site, Brandon, Florida
  - Research Site, Dunedin, Florida
  - Research Site, Largo, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Tampa, Florida
  - Research Site, Lawrenceville, Georgia
  - Research Site, Bowling Green, Kentucky
  - Research Site, Paducah, Kentucky
  - Research Site, Fall River, Massachusetts
  - Research Site, Battle Creek, Michigan
  - Research Site, Lincoln, Nebraska
  - Research Site, Smithtown, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Middleburg Heights, Ohio
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Hixson, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, Houston, Texas
  - Research Site, Victoria, Texas
  - Research Site, Chesapeake, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Clarksburg, West Virginia
- Canada (9):
  - Research Site, Victoria, British Columbia
  - Research Site, Quispamsis, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Burlington, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Research Site, Caguas, Puerto Rico

REFERENCES:
- [Background] Bessette L, Khraishi M, Kivitz AJ, Kaliyaperumal A, Grantab R, Poulin-Costello M, Isaila M, Collier D. Single-Arm Study of Etanercept in Adult Patients with Moderate to Severe Rheumatoid Arthritis Who Failed Adalimumab Treatment. Rheumatol Ther. 2017 Dec;4(2):391-404. doi: 10.1007/s40744-017-0079-x. Epub 2017 Sep 12. PMID 28900875
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 30 centers in the United States and Canada. Participants were enrolled from 06 May 2013 to 02 December 2014.
  Patients with moderate-to-severe rheumatoid arthritis (RA) who did not respond to or lost satisfactory response to adalimumab when used as the first biologic agent in combination with methotrexate were eligible.
Pre-assignment Details: A total of 90 participants were enrolled in the study, however, 4 participants from 1 site were excluded from all efficacy analyses due to good clinical practice (GCP) violations. Three of these participants who received etanercept are included in safety results.
Groups:
- Etanercept: Participants received 50 mg etanercept once weekly by subcutaneous injection with methotrexate for 24 weeks.
Period: Overall Study
Arm/Group | Etanercept
Started | 90
Received Etanercept | 88
Completed | 67
Not Completed | 23
Not completed — Withdrawal by Subject | 14
Not completed — Lost to Follow-up | 2
Not completed — Decision by Sponsor | 2
Not completed — Other | 1
Not completed — Ethical Reasons | 4

BASELINE CHARACTERISTICS:
Population: Full analysis set, which included all participants enrolled who received at least 1 dose of etanercept. Three additional participants were excluded from the FAS due to GCP violations.
Arm/Group | Etanercept
Number analyzed (Participants) | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 17
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Black (or African American) | 5
  Multiple | 1
  White | 74
  Other | 1
Anti-adalimumab Antibody Status [Number; unit: participants]
  Positive | 24
  Negative | 56
  Unknown | 5
Adalimumab Response Failure Type [Number; unit: participants] — Primary failure: Failure to achieve an American College of Rheumatology 20% improvement (ACR20) or equivalent as judged by the investigator; Secondary failure: Loss of an ACR20 response or equivalent as judged by the investigator.
  participants
    Primary | 33
    Secondary | 52

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 20 Response at Week 12
Description: A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 20% improvement in tender joint count; • ≥ 20% improvement in swollen joint count; and • ≥ 20% improvement in at least 3 of the 5 following parameters: o Patient Global Assessment of Joint Pain (measured on a 100 mm VAS); o Patient Global Assessment of Disease Activity (measured on a horizontal scale from 0 to 100); o Physician Global Assessment of Disease Activity (measured on a horizontal scale from 0 to 100); o Health Assessment Questionnaire - Disability Index (HAQ-DI) scale from 0 to 3, where zero represents no disability and three very severe, high-dependency disability; o C-reactive protein level.
Time Frame: Baseline and Week 12
Population: Full analysis set with non-missing data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 84
percentage of participants | 35.7 [25.6 to 46.9]

2. Secondary Outcome: Percentage of Participants With an ACR 20 Response at Week 12 by Anti-adalimumab Antibody Subgroup
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: Full analysis set with non-missing data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Presence of Anti-adalimumab Antibodies: Participants with anti-adalimumab antibodies.
- Absence of Anti-adalimumab Antibodies: Participants with absence of anti-adalimumab antibodies.
Arm/Group | Presence of Anti-adalimumab Antibodies | Absence of Anti-adalimumab Antibodies
Number analyzed (Participants) | 24 | 55
percentage of participants | 50.0 [29.1 to 70.9] | 32.7 [20.7 to 46.7]

3. Secondary Outcome: Percentage of Participants With an ACR 20 Response at Week 12 by Response Failure Type Subgroup
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: Full analysis set with non-missing data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Primary Failure: Participants failed to respond (defined as achievement of ACR20 or equivalent as judged by the investigator) to a combination treatment of adalimumab and methotrexate. This combination treatment must have been taken for at least 3 months.
- Secondary Failure: Participants who lost a satisfactory response (defined as achievement of ACR20 or equivalent as judged by the investigator) to a combination treatment of adalimumab and methotrexate. This combination treatment must have been taken for at least 6 months.
Arm/Group | Primary Failure | Secondary Failure
Number analyzed (Participants) | 33 | 51
percentage of participants | 27.3 [13.3 to 45.5] | 41.2 [27.6 to 55.8]

4. Secondary Outcome: Percentage of Participants With an ACR 20 Response at Week 24
Description: as for outcome 1
Time Frame: Baseline and Week 24
Population: Full analysis set with non-missing data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 84
percentage of participants | 34.5 [24.5 to 45.7]

5. Secondary Outcome: Percentage of Participants With an ACR 50 Response at Weeks 12 and 24
Description: A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 50% improvement in tender joint count; • ≥ 50% improvement in swollen joint count; and • ≥ 50% improvement in at least 3 of the 5 following parameters: o Patient Global Assessment of Joint Pain (measured on a 100 mm VAS); o Patient Global Assessment of Disease Activity (measured on a horizontal scale from 0 to 100); o Physician Global Assessment of Disease Activity (measured on a horizontal scale from 0 to 100); o Health Assessment Questionnaire - Disability Index (HAQ-DI) scale from 0 to 3, where zero represents no disability and three very severe, high-dependency disability; o C-reactive protein level.
Time Frame: Baseline and Weeks 12 and 24
Population: Full analysis set with non-missing data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 84
percentage of participants
  Week 12 | 10.7 [5.0 to 19.4]
  Week 24 | 15.5 [8.5 to 25.0]

6. Secondary Outcome: Percentage of Participants With an ACR 70 Response at Weeks 12 and 24
Description: A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 70% improvement in tender joint count; • ≥ 70% improvement in swollen joint count; and • ≥ 70% improvement in at least 3 of the 5 following parameters: o Patient Global Assessment of Joint Pain (measured on a 100 mm VAS); o Patient Global Assessment of Disease Activity (measured on a horizontal scale from 0 to 100); o Physician Global Assessment of Disease Activity (measured on a horizontal scale from 0 to 100); o Health Assessment Questionnaire - Disability Index (HAQ-DI) scale from 0 to 3, where zero represents no disability and three very severe, high-dependency disability; o C-reactive protein level.
Time Frame: Baseline and Weeks 12 and 24
Population: Full analysis set with non-missing data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 84
percentage of participants
  Week 12 | 2.4 [0.3 to 8.3]
  Week 24 | 3.6 [0.7 to 10.1]

7. Secondary Outcome: Change From Baseline in Disease Activity Score 28-C-Reactive Protein (DAS28-CRP)
Description: The DAS28-CRP is a composite score to measure disease activity in patients with rheumatoid arthritis, derived from the following variables:
  * The number of swollen and tender joints assessed using the 28-joint count;
  * C-reactive protein (CRP) level
  * Patient's global assessment of disease activity assessed on a score from 0 to 100.
  The DAS28-CRP score ranges from zero up to approximately ten. DAS28-CRP scores above 5.1 indicate high disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline and weeks 12 and 24
Population: Full analysis set, last observation carried forward imputation (LOCF) was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 84
units on a scale
  Week 12 | -1.10 (1.15)
  Week 24 | -1.33 (1.26)

8. Secondary Outcome: Percentage of Participants With DAS28-CRP Improvement of ≥ 1.2 Units From Baseline
Description: The DAS28-CRP is a composite score to measure disease activity in patients with rheumatoid arthritis, derived from the following variables: • The number of swollen and tender joints assessed using the 28-joint count; • C-reactive protein (CRP) level • Patient's global assessment of disease activity assessed on a score from 0 to 100. The DAS28-CRP score ranges from zero up to approximately ten. DAS28-CRP scores above 5.1 indicate high disease activity.
Time Frame: Baseline and weeks 12 and 24
Population: Full analysis set, last observation carried forward imputation (LOCF) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 84
percentage of participants
  Week 12 | 41.7 (1.15) [31.1 to 52.2]
  Week 24 | 48.8 (1.26) [38.1 to 59.5]

9. Secondary Outcome: Percentage of Participants With DAS 28-CRP < 3.2
Description: The DAS28-CRP is a composite score to measure disease activity in patients with rheumatoid arthritis, derived from the following variables: • The number of swollen and tender joints assessed using the 28-joint count; • C-reactive protein (CRP) level • Patient's global assessment of disease activity assessed on a score from 0 to 100. The DAS28-CRP score ranges from zero up to approximately ten. DAS28-CRP scores less than 3.2 are considered low disease activity.
Time Frame: Weeks 12 and 24
Population: Full analysis set, last observation carried forward imputation (LOCF) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 84
percentage of participants
  Week 12 | 13.1 (1.15) [5.9 to 20.3]
  Week 24 | 22.6 (1.26) [13.7 to 31.6]

10. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: The HAQ-DI is a questionnaire on which participants are asked to rate their level of difficulty on daily activities (dressing and grooming, arising, eating, and walking) and personal abilities (hygiene, reach, grip, and activity) as well as their use of aids, devices, or help from another person for these activities and disabilities. Responses are scored from 0 indicating no difficulty to 3 indicating inability to perform a task in that area. The overall score is the average of each of the 8 category scores and ranges from 0 (no disability) to 3 (very severe, high-dependency disability).
Time Frame: Baseline and weeks 12 and 24
Population: Full analysis set, last observation carried forward imputation (LOCF) was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 84
units on a scale
  Week 12 | -0.269 (0.540)
  Week 24 | -0.307 (0.602)

11. Secondary Outcome: Change From Baseline in 36-item Short Form Health Survey (SF-36) at Week 12
Description: The Medical Outcome Study Short Form 36-Item Health Survey, Version 2 (SF-36) is a self-administered instrument that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). Norm-based scores were used in analyses of each domain, calibrated so that 50 is the average score and the standard deviation equals 10. Higher scores indicate a higher level of functioning.
Time Frame: Baseline and Week 12
Population: Full analysis set; LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 82
units on a scale
  Physical Functioning | 4.46 (6.34)
  Role Physical | 3.34 (7.20)
  Bodily Pain | 4.27 (9.41)
  General Health | 2.86 (8.97)
  Vitality | 3.48 (9.31)
  Social Functioning | 3.06 (10.94)
  Role Emotional | 4.20 (9.80)
  Mental Health | 3.38 (9.24)

12. Secondary Outcome: Change From Baseline in 36-item Short Form Health Survey (SF-36) at Week 24
Description: as for outcome 11
Time Frame: Baseline and Week 24
Population: Full analysis set; LOCF imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 83
units on a scale
  Physical Functioning | 5.03 (7.66)
  Role Physical | 4.19 (7.68)
  Bodily Pain | 6.36 (9.72)
  General Health | 2.62 (8.64)
  Vitality | 4.65 (9.55)
  Social Functioning | 2.90 (10.42)
  Role Emotional | 4.49 (10.34)
  Mental Health | 3.66 (9.55)

13. Secondary Outcome: Work Productivity and Activity Impairment (WPAI)
Description: This 6-item assessment measures productivity losses during the past 7 days and includes measures on work time missed due to health, impairment while working due to health (the participant's assessment of the degree to which health affected their productivity while working), overall work impairment due to health (takes into account both hours missed due to health and the participant's assessment of the degree to which health affected their productivity while working) and activity impairment due to health (the degree in which health problems affected their ability to do regular daily activities). Scores for each measure are expressed from 0 to 100 with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes.
Time Frame: Baseline, week 12 and week 24
Population: Full analysis set participants who were employed (for the first 3 scores); LOCF imputation was used. "n" indicates the number of participants included in each analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 85
units on a scale
  Baseline: Percent Work Time Missed (n = 40) | 15.31 (27.76)
  Baseline: Percent Impairment While Working (n= 37) | 41.62 (24.44)
  Baseline: Percent Overall Work Impairment (n = 37) | 45.33 (26.36)
  Baseline: Percent Activity Impairment (n = 85) | 57.88 (21.77)
  Week 12: Percent Work Time Missed (n = 38) | 9.49 (24.85)
  Week 12: Percent Impairment While Working (n = 36) | 29.17 (23.59)
  Week 12: Percent Overall Work Impairment (n = 36) | 31.92 (25.57)
  Week 12: Percent Activity Impairment (n = 82) | 43.17 (24.99)
  Week 24: Percent Work Time Missed (n = 41) | 5.50 (17.71)
  Week 24: Percent Impairment While Working (n = 40) | 25.75 (23.74)
  Week 24: Percent Overall Work Impairment (n = 40) | 27.88 (24.79)
  Week 24: Percent Activity Impairment (n = 83) | 40.00 (26.82)

ADVERSE EVENTS:
Time Frame: 34 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 4/88
Other Adverse Events (participants affected / at risk) | 38/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=88)
Acute myocardial infarction (Cardiac disorders) | 1
Abdominal abscess (Infections and infestations) | 1
Cholecystitis infective (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Altered state of consciousness (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=88)
Nausea (Gastrointestinal disorders) | 7
Injection site erythema (General disorders) | 7
Injection site reaction (General disorders) | 6
Bronchitis (Infections and infestations) | 6
Sinusitis (Infections and infestations) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 5
Headache (Nervous system disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.